CLINICAL TRIAL: NCT00890058
Title: A Case Control Study to Define Clinical, Immunologic and Radiographic Features of the Aromatase Inhibitor Arthralgia Syndrome
Acronym: CIRAS
Status: Completed | Type: Observational
Sponsor: Victoria Shanmugam (Other)
Responsible Party: Sponsor-Investigator, Victoria Shanmugam, Associate Professor of Medicine, George Washington University
Organization: George Washington University (Other)
Other Study IDs: 2008-547
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Arthralgia Syndrome; Arthritis; Synovitis
Keywords: Arthritis; Synovitis; Aromatase Inhibitor; Arthralgia Syndrome
MeSH Terms: conditions — Arthritis; Synovitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for cytokine measurements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Postmenopausal breast cancer patients with hand pain receiving aromatase inhibitors
- Controls: Postmenopausal breast cancer patients with hand pain not receiving aromatase inhibitors

SUMMARY:
The CIRAS study will investigate postmenopausal breast cancer patients with hand pain and compare those receiving aromatase inhibitors (cases) to breast cancer patients with hand pain not receiving aromatase inhibitors (controls) in order assess whether this syndrome is an inflammatory arthritis.

DETAILED DESCRIPTION:
This study is for women with post-menopausal breast cancer and hand pain. Patients do not need to be taking aromatase inhibitors to be eligible for the study. We want to study the joint findings in patients with hand pain and breast cancer undergoing treatment with aromatase inhibitor medications and compare them to patients with hand pain and breast cancer not treated with these medications.

Aromatase inhibitor drugs are used in certain types of breast cancer to reduce the risk of cancer returning after treatment. One of the side effects of aromatase inhibitors is the development of joint pain, a complication known as the Arthralgia Syndrome. The cause of the Arthralgia Syndrome is not known, but we suspect that the pain may be due to inflammation in the joints. Currently, the only effective treatment is to stop the aromatase inhibitor, and so affected patients may miss out on an otherwise useful treatment to prevent return of their cancer.

Post-menopausal patients with breast cancer and hand pain can enroll in the study. Patients will be asked to come for a separate visit which will take about half a day.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged over 18 with stage I-III breast cancer undergoing treatment at the Lombardi Cancer Center.
2. Presence of hand pain
3. No active signs of ongoing malignant disease

Exclusion Criteria:

1. Known autoimmune disease for example, rheumatoid arthritis, systemic lupus erythematosis, polymyalgia rheumatica, or seronegative arthritis.
2. Age <18
3. Unable to complete informed consent process

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with stage I-III breast cancer currently undergoing treatment at the Lombardi Cancer Center will be screened for the presence of joint and hand symptoms.Patients with symptoms who are receiving aromatase inhibitors will be considered to be cases, while those with symptoms who are not receiving aromatase inhibitors will be considered to be controls.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Difference in DAS-28 between cases and controls | 1 year

SECONDARY OUTCOMES:
Differences between cases and controls in mean ESR, TNF-alpha, IL-6 and ultrasound measurement of tenosynovitis. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Shanmugam, MD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Shanmugam VK, McCloskey J, Elston B, Allison SJ, Eng-Wong J. The CIRAS study: a case control study to define the clinical, immunologic, and radiographic features of aromatase inhibitor-induced musculoskeletal symptoms. Breast Cancer Res Treat. 2012 Jan;131(2):699-708. doi: 10.1007/s10549-011-1849-8. Epub 2011 Nov 11. PMID 22076476